CLINICAL TRIAL: NCT01298310
Title: A Randomised, Double-blind, Placebo-controlled, Three-way Cross-over Single Center Study to Characterize the Phenotype in Patients With Morton's Neuroma and to Explore the Effect of Local Administration of Xylocaine (Lidocaine)
Brief Title: A Study to Characterize the Phenotype in Patients With Morton's Neuroma and to Explore the Effect of Local Administration of Xylocaine (Lidocaine)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: D2285M00032; Eudract no: 2010-024295-26
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Morton's Neuroma
Keywords: Morton's neuroma, QST measurements
MeSH Terms: conditions — Morton Neuroma | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Xylocaine_1mg (Active Comparator): 1 injection of Xylocaine (1 mg/mL)
  Interventions: Drug: Xylocaine
- Xylocaine_10mg (Active Comparator): 1 injection of Xylocaine (10 mg/mL)
  Interventions: Drug: Xylocaine
- Placebo (Placebo Comparator): 1 injection of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xylocaine — 1 mg/mL solution for injection
  Arms: Xylocaine_1mg
Drug: Xylocaine — 10 mg/mL solution for injection
  Arms: Xylocaine_10mg
Drug: Placebo — solution for injection
  Arms: Placebo

SUMMARY:
To characterize the phenotype in patients with Morton's neuroma and to explore the effect of local administration of Xylocaine (lidocaine)

DETAILED DESCRIPTION:
A randomised, double-blind, placebo-controlled, three-way cross-over single center study to characterize the phenotype in patients with Morton's Neuroma and to explore the effect of local administration of Xylocaine (lidocaine)

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of Morton's neuroma with symptoms of at least 3 months duration in one foot (affected foot)
* Visual analogue scale (VAS) pain-score of = 40 mm in the painful foot at daily activities during the previous week (visit 1)

Exclusion Criteria:

* Allergy to lidocaine
* Scars or other dermal conditions on the feet that may interfere with study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The baseline phenotypic Quantitative sensory testing (QST) variables (e.g. heat, cold, touch and mechanical pain perception). Sensory tests will be performed to measure pain and skin sensitivity by use of different pressure (mN) and temperature ( C) | Before and after drug injection at Day 1
The baseline phenotypic Quantitative sensory testing (QST) variables (e.g. heat, cold, touch and mechanical pain perception). Sensory tests will be performed to measure pain and skin sensitivity by use of different pressure (mN) and temperature ( C) | Before and after drug injection at Day 14 (+/-9).
The baseline phenotypic Quantitative sensory testing (QST) variables (e.g. heat, cold, touch and mechanical pain perception). Sensory tests will be performed to measure pain and skin sensitivity by use of different pressure (mN) and temperature ( C) | Before and after drug injection at Day 28 (+/-18).
The effect of Xylocaine compared to placebo in QST variables. Sensory tests will be performed to measure pain and skin sensitivity by use of different pressure (mN) and temperature ( C) | After drug injection at Day 1.
The effect of Xylocaine compared to placebo in QST variables. Sensory tests will be performed to measure pain and skin sensitivity by use of different pressure (mN) and temperature ( C) | After drug injection at Day 14 (+/-9).
The effect of Xylocaine compared to placebo in QST variables. Sensory tests will be performed to measure pain and skin sensitivity by use of different pressure (mN) and temperature ( C) | After drug injection at Day 28 (+/-18).

SECONDARY OUTCOMES:
Frequency/severity of adverse events | Day 1
Frequency/severity of adverse events | Day 14 (+/-9)
Frequency/severity of adverse events | Day 28 (+/-18)
Frequency/severity of adverse events | Day 43 (+/-32)

CONTACTS AND LOCATIONS:
Overall Officials: Bror Jonzon, MD, PhD, Study Director — AstraZeneca R&D Södertälje, Sweden
Locations (1):
- Research Site, Stockholm, Sweden